CLINICAL TRIAL: NCT03593486
Title: Effect of Low-Level Electromagnetic Field Stimulation on Patients With Paroxysmal Atrial Fibrillation
Brief Title: Low-Level EMF Stimulation for Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMF for Atrial Fibrillation
Record Dates: First submitted 2018-06-24; First posted 2018-07-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Autonomic Imbalance
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to either the active or sham stimulation group. Because the parameters are programmed into the stimulator by the manufacturer and given generic names (Stim 1 and Stim 2), the investigators and physicians performing the procedure will not know which protocol is active or sham.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Stimulation (Experimental): Participants will receive active EMF stimulation through the study device for 60 minutes during the procedure.
  Interventions: Device: Low-level Pulsed EMF
- Sham Stimulation (Sham Comparator): The participant will be positioned in the stimulator, but no EMF stimulation will be delivered.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Low-level Pulsed EMF — Low-level pulsed electromagnetic field stimulator delivered through a Helmholtz coil positioned around the participant's head and neck. Stimulation parameters are 0.032 µG at 0.89 Hz for 60 minutes.
  Arms: Active Stimulation
Device: Sham Stimulation — The stimulator will be placed around the participant's head and neck, but no EMF will be delivered.
  Arms: Sham Stimulation

SUMMARY:
This research has two main specific aims. First, a commercially-available stimulator will be utilized to assess the effect of low-level electromagnetic field (EMF) stimulation on atrial fibrillation (AF) inducibility in patients with paroxysmal AF presenting for catheter ablation as compared to sham stimulation. We hypothesize a reduction in AF inducibility in patients treated with EMF stimulation. Second, we aim to assess for the effect of low-level EMF on level of systemic inflammatory mediators. We hypothesize a reduction in the level of the inflammatory mediator tissue necrosis factor (TNF)-α in patients treated with EMF stimulation as compared to sham stimulation. The long-term objective of this research is to develop low-level EMF as a therapeutic alternative for patients with AF, and this research will help to determine the efficacy of low-level pulsed EMF in this regard.

DETAILED DESCRIPTION:
This is a prospective, randomized, sham-controlled trial. Patients will be enrolled upon presentation to our electrophysiology (EP) lab for ablation of paroxysmal AF. After informed consent is obtained, the patient will be randomized to one of two protocols that have been pre-programmed into the magnetic field stimulator. As described below, one of the protocols will be an active stimulation protocol, and one will be sham (i.e. no stimulation delivered). These will be named "Stim 1" and "Stim 2" in the computer. Because the specifics of the protocol are programmed into the stimulator by the device manufacturer, investigators will not know which of these two protocols is active vs. sham. The patient will then be brought to the EP lab for the procedure and will be placed on the lab table with their head positioned in the magnetic coil. Vascular access will then be obtained and diagnostic catheters placed as is standard practice for AF ablation.

Because the study is limited to patients with paroxysmal AF, patients will begin the study in normal sinus rhythm (NSR). Before the experimental protocol is begun, baseline electrophysiologic intervals will be recorded as is standard practice for all patients presenting for EP study. This will include measurement of the atrio-ventricular nodal effective refractory period (AVNERP) using programmed stimulation from the right atrial (RA) appendage, atrio-his (AH) interval, and his-ventricular (HV) interval per standard practice. Burst atrial pacing will then be utilized to induce AF. Measurements of the number of burst pacing attempts required to induce AF, as well as the AF cycle length, and duration of pacing-induced AF will be recorded. Attempts at AF induction will occur for 15 minutes. Prior to induction of AF, 5ml of venous blood will be drawn from the central venous sheaths to measure baseline levels of the inflammatory mediator (TNF)-α. These samples will be stored for analysis.

After baseline measurements are obtained, the coil will be turned on and whichever protocol the patient has been assigned to will be run. The system to be used contains a signal-generator coupled to a Helmholtz coil capable of producing a magnetic field in response to an electric current. The Helmholtz coil itself is has 9 inches of separation in between the two coils that allows for placement of the coil around the participant's head and upper neck. The choice of the head and neck as the site of stimulation is intended to target the vagus nerve as it exits the jugular foramen to course caudally in the carotid sheath. The system is designed to create a homogenous, isotropic magnetic field with a field strength from 1 to 99 pico-Tesla (pT) with a frequency range of 0.01 Hz to 50 Hz.

Active Stimulation will involve application of a pulsed-EMF with the parameters 0.032 micro-gauss (µG) at 0.89 Hz for 60 minutes. In participants randomized to sham stimulation, the coil will be positioned around the neck as previously described, but no current will be applied to the stimulator.

During the 60 minute stimulation time, trans-septal puncture and mapping of the left atrium will be performed as is standard practice for this procedure, but no ablation will be performed. After the 60 minute protocol is complete, venous blood samples will again be drawn (within 5 minutes of protocol completion), stored, and analyzed as previously described. If the patient remains in AF after the end of the 60 minute session, they will be electrically cardioverted to sinus rhythm. The same stimulation protocol as described previously will again be employed, again noting number of attempts required to induce AF, duration of pacing-induced AF, AF cycle length, and measurements of AVNERP, AH, HV intervals and levels of TNF-α.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21-85 presenting for ablation of paroxysmal atrial fibrillation (episodes of atrial fibrillation lasting < 7 days with or without prior cardioversion)

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 40%
* Stroke or myocardial infarction within the past 6 months
* Greater than moderate valvular stenosis or regurgitation as assessed by pre-procedure transthoracic echocardiogram (TTE)
* Presence of a prosthetic heart valve.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Change in duration of pacing-induced atrial fibrillation | 60 minutes
  Change in the duration of atrial fibrillation that is induced by burst-pacing compared between the two groups before and after the stimulation period.

SECONDARY OUTCOMES:
Number of pacing attempts required to induce AF | 60 minutes
  Number of burst-pacing attempts that are required to successfully induced atrial fibrillation, compared between the two groups before and after the stimulation period.
AF Cycle length | 60 minutes
  Cycle length of induced atrial fibrillation, compared between the two groups before and after the stimulation period.
TNF-alpha levels | 60 minutes
  Levels of the inflammatory mediator TNF-alpha measured in central venous blood, compared between the two groups before and after the stimulation period.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Po, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Zhou X, Wang Z, Huang B, Zhou L, Chen M, Yu L, Jiang H. Magnetic fields in noninvasive heart stimulation: A novel approach for anti-atrial fibrillation. Int J Cardiol. 2015;190:54-5. doi: 10.1016/j.ijcard.2015.04.155. Epub 2015 Apr 21. No abstract available. PMID 25912123
- [Background] Chen PS, Chen LS, Fishbein MC, Lin SF, Nattel S. Role of the autonomic nervous system in atrial fibrillation: pathophysiology and therapy. Circ Res. 2014 Apr 25;114(9):1500-15. doi: 10.1161/CIRCRESAHA.114.303772. PMID 24763467
- [Background] Scherlag BJ, Yamanashi WS, Hou Y, Jacobson JI, Jackman WM, Lazzara R. Magnetism and cardiac arrhythmias. Cardiol Rev. 2004 Mar-Apr;12(2):85-96. doi: 10.1097/01.crd.0000094029.10223.2f. PMID 14766023
- [Background] Yu L, Dyer JW, Scherlag BJ, Stavrakis S, Sha Y, Sheng X, Garabelli P, Jacobson J, Po SS. The use of low-level electromagnetic fields to suppress atrial fibrillation. Heart Rhythm. 2015 Apr;12(4):809-17. doi: 10.1016/j.hrthm.2014.12.022. Epub 2014 Dec 19. PMID 25533588
- [Background] Stavrakis S, Humphrey MB, Scherlag BJ, Hu Y, Jackman WM, Nakagawa H, Lockwood D, Lazzara R, Po SS. Low-level transcutaneous electrical vagus nerve stimulation suppresses atrial fibrillation. J Am Coll Cardiol. 2015 Mar 10;65(9):867-75. doi: 10.1016/j.jacc.2014.12.026. PMID 25744003